CLINICAL TRIAL: NCT06179862
Title: Effects of Hamstring Shortness on Jump Performance in Young Basketball Players Impact
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: E-85646034-604.02.02-67240
Record Dates: First submitted 2023-12-08; First posted 2023-12-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Hamstring Injury
Keywords: basketball; shortness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the realm of sports performance, particularly in disciplines demanding explosive lower-body strength and agility, such as basketball, an athlete's ability to execute powerful and high-reaching jumps plays a pivotal role. Optimal lower-extremity flexibility, particularly in the hamstrings, is crucial for achieving maximum vertical jump height. Hamstring shortness, characterized by limited flexibility and reduced muscle extensibility, is frequently observed among athletes and has been linked to compromised jump performance.

DETAILED DESCRIPTION:
Young basketball players, in their developmental stages, often face the challenge of balancing strength, flexibility, and functional movement. Hamstring tightness is a prevalent issue among this demographic, potentially influencing their ability to generate adequate power during jumps. The impact of hamstring shortness on jump performance is multifaceted, affecting the force production, range of motion, and efficiency of movement crucial for executing explosive jumps

ELIGIBILITY:
Inclusion criteria

* To be between 10-16 years old
* Being a licensed basketball player
* Playing in the Istanbul Local Basketball League run by the Turkish Basketball Federation
* Sit-to-Face test 30 cm and below Goniometric measurement less than 80 degrees in active straight leg raising test, Exclusion criteria
* Having played one match in the 48 hours prior to the evaluation
* Having a lower extremity injury.
* Participants of both genders will be included in the study.

Ages: 10 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Amateur basketball players will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Goniometric Measurement | day 1
  The individual who will participate in the evaluation is placed in the supine position. After taking the ankle of the participant's leg, which we will measure, to neutral, the participant passively flexes the leg at the hip. When the participant feels resistance during this movement, when pain sensation occurs and at the last point where the knee starts to bend, the measurement is taken with a goniometer. In the goniometric measurement, the pivot point is based on the trochanter major and the fixed arm is parallel to the trunk. If a value below 80 degrees is obtained as a result of the measurement, it is seen that hamstring shortness is present in this person.
sit and reach | day 1
  Individuals who will participate in the assessment are asked to remove their shoes and socks. The individuals to be evaluated sit in a long sitting position with the soles of their feet in full contact with the measuring board. The participant is asked to push the iron bar by slowly reaching towards his/her toes with both hands without bending his/her knees. The point on the pushed bar where the individual can reach the maximum distance without bending his/her knees is taken as a criterion. If the iron bar is below 30 cm, it shows that the hamstring muscle is short and the test is positive
Y Balance Test | day 1
  In order to apply the Y balance test, a large letter Y is taped to the ground on a flat surface so that the angle between the front and back directions is 135 degrees and the angle between the two back sides is 90 degrees. The participant to be tested is asked to move to the center of the line. The participant is instructed that while balancing on one foot, he/she should reach anteriorly, posterolaterally and posteromedially with the other foot and keep his/her weight on the stable foot. . For score calculation, the distance lengths in three directions obtained with the participant's previously measured leg length are summed, divided by 3 times and multiplied by 100 to obtain the score
Popliteal Angle Measurement (Holt Method) | day 1
  While the person to be evaluated is lying on his/her back, the knee and hip are flexed 90 degrees. After assuming this position, the individual is asked to extend the knee until a resistance is encountered. The angle between the vertical axis of the knee and the last point reached in the movement is measured and this angle is expected to be 0-10 degrees in normal individuals. If full extension cannot be performed, hamstring shortness is determined
vertical jump Height | day 1
  The optojump system will be used in this study as a jumping power measurement tool.
  In the measurements, the vertical jump height was recorded with the optoJump system and the software of this system (Microgate, Bolzano, Italy). The measurement of the vertical jump distance in centimeters is done by means of two bars in the OptoJump system with sensors that detect movement.
The duration of the jump (milliseconds) | day 1
  The optojump system will be used in this study as a jumping power measurement tool.
  The duration of the jump (milliseconds) is also included in determining the jump distance.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)